CLINICAL TRIAL: NCT05959148
Title: Would Integrating Monochromatic Infrared Energy Into the Physical Rehabilitation of Adolescents With Patellofemoral Pain Syndrome Have Any Advantageous Effects? a Randomized Controlled Trial
Brief Title: Adjuvant Effects of Monochromatic Infrared Energy in Rehabilitation of Adolescents With Patellofemoral Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ragab Kamal Elnaggar, Associate Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHPT/0021/0026
Record Dates: First submitted 2023-07-15; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Intervention Model Description: A prospective, randomized controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: This was a single-blind protocol. The outcome assessor was blinded to the treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIRE group (Experimental): Participants in this group underwent MIRE application in addition to the traditional physical therapy program
  Interventions: Other: Monochromatic infrared energy
- Control (Active Comparator): Participants in this group received the traditional physical therapy program only.
  Interventions: Other: Traditional physical therapy

INTERVENTIONS:
Other: Monochromatic infrared energy — The monochromatic infrared energy was delivered through an Anodyne Therapy Professional Infrared Therapy System. Light energy (parameter: a wavelength of 890 nm and radiant power at a rate of 6.24 W) was produced through 8 array diode therapy pads applied on both knees (on the medial, lateral, anterior, and posterior aspects of each knee), each including 60 super-luminescent gallium-aluminum arsenide diodes. The MIRE was applied for 40 minutes/session, three times a week, for three successive months.
  Arms: MIRE group
Other: Traditional physical therapy — The traditional physical therapy program consisted of stretching and strengthening exercises for the muscles surrounding the hip and knee, balance exercises, as well as other electrotherapeutic modalities (ultrasound and hot application).
  Arms: Control

SUMMARY:
This study assessed if integrating monochromatic infrared energy (MIRE) would affect pain, dynamic postural control, functional status, and health-related quality of life in adolescents with patellofemoral pain syndrome (PFPS). Forty-six patients with PFPS were randomly allocated to the MIRE group (n = 23, received the received MIRE in addition to the traditional physical therapy program) or the control group (n = 23, received the traditional physical therapy program only). Both groups were assessed for pain, dynamic postural control, functional status, and health-related quality before and after intervention.

DETAILED DESCRIPTION:
Forty-six adolescents with PFPS were recruited from the university's outpatient orthopedic and physical therapy clinics and two referral hospitals in AlKharj, Saudi Arabia. The study included patients who were 15-18 years old, had anterior-knee or retro-patellar pain that increase with activities like squatting, running, prolonged sitting, or stair climbing, had PFPS with insidious onset for more than 6 weeks without any traumatic incidence, and were not participating in a regular exercise program in the past 3 months. Patients who had meniscal tears, collateral/cruciate ligament injury, knee arthritis, a history of knee/hip surgery, or previous patellar subluxation/dislocation were excluded.

Outcome measures

Pain: Pain during rest and/or movement was assessed using the Numerical Pain Rating Scale.

Dynamic postural control: The dynamic postural control was assessed through the modified star excursion balance test (mSEBT).

Functional status: The functional status was evaluated using the Arabic version of the Anterior Knee Pain Questionnaire (Kujala Questionnaire).

Quality of life: The quality of life was assessed through the self-report Pediatric Quality of Life Inventory.

Interventions

The MIRE group underwent MIRE application on the affected knee for 40 minutes, 3 times a week for 3 consecutive months. The MIRE was delivered using an Anodyne Therapy Professional Infrared Therapy System (parameter: a wavelength of 890 nm and radiant power at a rate of 6.24 W). Participants in the MIRE group further received the traditional physical therapy program (60 minutes/session) that consisted of stretching and strengthening exercises for the muscles surrounding the hip and knee, balance exercises, as well as other electrotherapeutic modalities (ultrasound and hot application). The control group received the traditional physical therapy program only.

ELIGIBILITY:
Inclusion Criteria:

* Age between15 and18 years.
* Anterior-knee or retro-patellar pain that increases with activities like squatting, running, prolonged sitting, or stair climbing.
* PFPS with insidious onset for more than 6 weeks without any traumatic incidence.
* Not participating in a regular exercise program within the last three months.

Exclusion Criteria:

* Meniscal tears
* Collateral/cruciate ligament injury
* Knee arthritis
* History of hip/knee surgery
* Previous patellar subluxation/dislocation

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2021-10-03 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-09-29 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 3 months
  Participants reported how much they feel pain during rest and/or movement on the 0-10 Visual Analogue Scale, where 0 represents "no pain" and 10 indicates the "worst possible pain".
Dynamic postural control | 3 months
  The dynamic postural control was assessed through the modified star excursion balance test (mSEBT). Participants stood in the middle of a floor grid with three reach lines creating a Y shape. They were told to stand on one limb and extend as far as they could with the distal end of the reaching limb pointed in each anterior, posteromedial, and posterolateral direction. The distance from the center to the point of the foot reach was then measured with a measuring tape (in/cm), and the reaching limb was restored to the starting position. The composite reach distance of the three directions was calculated and normalized to the length of the leg and used for data analysis. The higher the normalized mSEBT score the better the postural control.

SECONDARY OUTCOMES:
Functional status | 3 months
  To evaluate functional status, the Arabic version of the Anterior Knee Pain Questionnaire (Kujala Questionnaire) was utilized. It measures the functional limitations imposed on by patellofemoral pain with 13 self-reported items. Six physical activities-sitting, squatting, walking, climbing stairs, leaping, and running-were chosen to assess pain, abnormal patellar movement, edema, limited knee flexion, and quadriceps atrophy. The score is 0 to 100, with 100 representing no discomfort or functional impairment and 0 representing total functional incapacity.
Life quality | 3 months
  To evaluate the quality of life, the self-report Pediatric Quality of Life Inventory (PedsQL) was utilized. It is a 23-item multidimensional assessment of children's and adolescents' health-related quality of life that is broken down into four domains: physical (8 items), emotional (5 items), social (5 items), and school-related (3 items). Scores range from 0 (never) to 4 (almost always) for each item. The scale for the items is linear reversed on a 0-100 scale, with 0=100, 1=75, 2=50, 3=25, and 4=0. Higher scores denotes better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ragab K. Elnaggar, PhD, Principal Investigator — Prince Sattam Bin Abdulaziz University
Locations (1):
- Ragab K. Elnaggar, Al Kharj, Riyadh Region, Saudi Arabia